CLINICAL TRIAL: NCT00542165
Title: Multicenter Prospective Study on the Changes of Sexual Function Following Treatment With Alfuzosin (Xatral XL) in Patients With Benign Prostatic Hypertrophy
Brief Title: Multicenter Prospective Study on the Changes of Sexual Function Following Treatment With Alfuzosin (Xatral XL®) in Patients With Benign Prostate Hypertrophy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L_8819
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: BPH/LUTS/Sexual Functions
MeSH Terms: interventions — alfuzosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfuzosin

SUMMARY:
To collect under daily practice conditions, clinical data on the changes of sexual function when a new formulation of alfuzosin(Xatral XL® )is administered once daily in patients with lower urinary tract symptoms(LUTS) suggestive of prostatic hypertrophy

ELIGIBILITY:
Inclusion Criteria:

* male patients suffering from LUTS lasting 6months and over
* male patients aged 50 years old and over who has a continuous active partner

Exclusion Criteria:

* Primary hypogonadism and neuropathy patients
* History of prostate surgery
* Patients with prostate cancer
* History of organ surgery or organ damage in pelvis
* History of myocardiac infarction, stroke, and life threatening arrythmia within last 6 months
* Patients with haematuria caused by other reasons except BPH
* Patients with uncontrolled hypertension in spite of treatment with antihypertensive agents
* History of a malignant tumor within last 5 years
* Patients who are currently controlled with other medication for erectile dysfunction
* Patients who have been administered with androgen or antiandrogen
* Patients who is treated for psychiatric disorder or depression
* Combination with other alpha1-blockers
* Patients previously not improved by an alpha1-blocker treatment
* Known hypersensitivity to the alfuzosin
* History of postural hypotension or syncope
* Hepatic insufficiency
* Unstable angina pectoris

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2004-03; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
IIEF and GEQ (Global Efficacy Question) | at intermediate visit (M1) and at end-point visit(M3)

SECONDARY OUTCOMES:
blood pressure and heart rate measure in sitting position | at each visit
IPSS and Quality of Life Score | at intermediate visit (M1) and at end-point visit(M3)
Maximum flow rate and post voiding residual urine | at end-point visit(M3)
Spontaneous reported adverse events | During all the study period

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Young Ahn, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Seoul, South Korea